CLINICAL TRIAL: NCT02590263
Title: A Non-Randomized, Open-Label, Multi-Center Phase 1/2 Study Evaluating the Safety, Pharmacokinetics and Efficacy of ABT-414 in Japanese Subjects With Malignant Glioma
Brief Title: Study Evaluating ABT-414 in Japanese Subjects With Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-714
Record Dates: First submitted 2015-09-28; First posted 2015-10-29 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Malignant Glioma; Glioblastoma Multiforme
Keywords: WHO grade III; WHO grade IV; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma; Lymphoma, Follicular | interventions — Temozolomide; ABT-414; depatuxizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A of Phase 1 portion (Experimental): ABT-414 administered every other weeks monotherapy
  Interventions: Drug: ABT-414
- Phase 2 portion (Experimental): ABT-414 administered every other weeks in combination with temozolomide
  Interventions: Drug: Temozolomide; Drug: ABT-414
- Arm C of Phase 1 portion (Experimental): ABT-414 administered every other weeks in combination with radiation and temozolomide
  Interventions: Radiation: Whole Brain Radiation; Drug: Temozolomide; Drug: ABT-414
- Arm B of Phase 1 portion (Experimental): ABT-414 administered every other weeks in combination with radiation and temozolomide
  Interventions: Radiation: Whole Brain Radiation; Drug: Temozolomide; Drug: ABT-414

INTERVENTIONS:
Radiation: Whole Brain Radiation — Whole Brain Radiation will be administered in over 30 fractions as per the procedure in each study site.
  Arms: Arm B of Phase 1 portion; Arm C of Phase 1 portion
Drug: Temozolomide — Temozolomide will be administered per label.
  Arms: Arm B of Phase 1 portion; Arm C of Phase 1 portion; Phase 2 portion
Drug: ABT-414 — ABT-414 will be administered by intravenous infusion
  Other Names: Depatuxizumab; Mafodotin

SUMMARY:
This study seeks to evaluate the tolerability, pharmacokinetics (PK), efficacy, and safety of ABT-414 in Japanese participants with newly diagnosed and recurrent, World Health Organization (WHO) grade III or IV malignant glioma.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants with WHO grade III or IV malignant glioma
* 70 or above on Karnofsky Performance Status in Arm A of Phase 1 portion and Phase 2 portion
* 80 or above on Karnofsky Performance Status in Arm B and Arm C of Phase 1 portion
* Adequate bone marrow function
* Recurrent malignant glioma per RANO criteria in Arm A of Phase 1 portion and Phase 2 portion
* Histologically proven newly diagnosed malignant glioma in Arm B and Arm C of Phase 1 portion
* Participants must have confirmed EGFR amplification by central lab in Phase 2 portion

Exclusion Criteria:

* Anti-cancer treatment 28 days prior to study Day 1 for Arm A of Phase 1 portion and Phase 2 portion (except temozolomide therapy for newly diagnosed treatment for Phase 2 portion)
* Anti-cancer treatment prior to study Day 1 for Arm B and Arm C of Phase 1 portion
* Participant has received prior treatment with bevacizumabor, EGFR therapy in Arm A of Phase 1 portion and Phase 2 portion, or for recurrent glioblastoma in Phase 2 portion
* Participant has a history of major immunologic reaction to any Immunoglobulin G containing agents or component of ABT-414.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events | At each visit for approximately 4 years
Number of Dose Limiting Toxicities | At each visit for approximately 1 year
  Measurement by clinical lab results, vital signs, physical exam and electrocardiogram (ECG) during the Phase 1 portion of the study.
Progression-free survival | At each visit for approximately 1 year
  Time to progression-free survival is defined as the number of days from the date of first dose to the date of earliest disease progression based on Response Assessment in Neuro-Oncology (RANO) criteria or to the date of death, if disease progression does not occur (except Arm B and Arm C of Phase 1 portion).
Area under the plasma concentration-time curve (AUC) of ABT-414 | Multiple time points in Cycles 1, 2 and 3 (4 weeks each) and Day 1 of remaining cycles until end of treatment for approximately 1 year for recurrent subjects and in every week of Day 1 until Week 7 and end of treatment for the newly diagnosed subjects
  Assessed during the Phase 1 portion of the study, the area under the plasma concentration-time curve (AUC) is a method of measurement to determine the total exposure of a drug in blood plasma.
Maximum plasma concentration (Cmax) of ABT-414 | Multiple time points in Cycles 1, 2 and 3 (4 weeks each) and Day 1 of remaining cycles until end of treatment for approximately 1 year for recurrent subjects and in every week of Day 1 until Week 7 and end of treatment for the newly diagnosed subjects
  Assessed during the Phase 1 portion of the study, the maximum plasma concentration (Cmax) is the highest concentration that a drug achieves in the blood after administration in a dosing interval.

SECONDARY OUTCOMES:
Objective Response Rate | At each visit for approximately 1 year
  The objective response rate is defined as the proportion of participants with at least one measurable lesion at baseline who achieves a confirmed complete (CR) or partial response (PR) based on RANO criteria (except Arm B and Arm C of Phase 1 portion).
Overall Survival | At each visit for approximately 1 year
  Overall survival is defined as number of days from the date of first dose to the date of death for all dosed participants (except Arm B and Arm C of Phase 1 portion).
Duration of Overall Response | At each visit for approximately 1 year
  The duration of overall response for a given participant is defined as the number of days from the day the RANO criteria are met for CR or PR (whichever is recorded first) to the date that progressive disease (PD) is objectively documented (based RANO criteria) (except Arm B and Arm C of Phase 1 portion).

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (22):
- Japan (22):
  - Nagoya University Hospital /ID# 138559, Nagoya, Aichi-ken
  - Hiroshima University Hospital /ID# 139399, Hiroshima, Hiroshima
  - Hokkaido University Hospital /ID# 150589, Sapporo, Hokkaido
  - University of Tsukuba Hospital /ID# 140433, Tsukuba, Ibaraki
  - Iwate Medical University Hospital /ID# 149145, Shiwa-gun, Iwate
  - Kitasato University Hospital /ID# 148493, Sagamihara-shi, Kanagawa
  - Kumamoto University Hospital /ID# 138558, Kumamoto, Kumamoto
  - Kyoto Prefect Univ Med /ID# 149093, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 163206, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 138464, Sendai, Miyagi
  - Okayama University Hospital /ID# 148674, Okayama, Okayama-ken
  - Osaka University Hospital /ID# 140438, Suita-shi, Osaka
  - Saitama Medical University International Medical Center /ID# 140361, Hidaka-shi, Saitama
  - Shizuoka Cancer Center /ID# 148673, Sunto-gun, Shizuoka
  - Dokkyo Medical University Hospital /ID# 150990, Shimotsuga-gun, Tochigi
  - National Cancer Center Hospital /ID# 140435, Chuo-ku, Tokyo
  - Nihon University Itabashi Hospital /ID# 149385, Itabashi-ku, Tokyo
  - Kyorin University Hospital /ID# 140360, Mitaka-shi, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 140436, Shinjuku-ku, Tokyo
  - Chiba Cancer Center /ID# 164375, Chiba
  - NHO Kyoto Medical Center /ID# 140437, Kyoto
  - Osaka International Cancer Institute /ID# 148494, Osaka

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Narita Y, Muragaki Y, Kagawa N, Asai K, Nagane M, Matsuda M, Ueki K, Kuroda J, Date I, Kobayashi H, Kumabe T, Beppu T, Kanamori M, Kasai S, Nishimura Y, Xiong H, Ocampo C, Yamada M, Mishima K. Safety and efficacy of depatuxizumab mafodotin in Japanese patients with malignant glioma: A nonrandomized, phase 1/2 trial. Cancer Sci. 2021 Dec;112(12):5020-5033. doi: 10.1111/cas.15153. Epub 2021 Oct 30. PMID 34609773